CLINICAL TRIAL: NCT01100593
Title: Optimal Catheter Length for Ultrasound-Guided Peripheral Vascular Access
Brief Title: Ultrasound IV Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 28195
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: IV Access; Ultrasound Use
Keywords: Ultrasound; IV catheters; Extravasation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.75 inch catheter length (Active Comparator): Length of catheter to be used
  Interventions: Procedure: length of IV catheter
- 2.5 inch catheter length (Active Comparator): length of catheter to be used
  Interventions: Procedure: length of IV catheter

INTERVENTIONS:
Procedure: length of IV catheter — Subjects will be randomized to one of two IV catheter lengths

SUMMARY:
The purpose of this study is to compare catheter length and extravasation rates for Ultrasound (US)-guided peripheral intravenous (IV) catheter insertion in a subset of emergency department patients with difficult IV access. Physicians, Emergency RNs, and Emergency Technicians can be taught to use US guidance to start peripheral IV in the ED. The optimal length of catheter to use for this procedure is unknown. This study will provide data on the length of catheter required to minimize extravasation. There is no guideline on catheter length selection for US-guided peripheral vascular access. This study may decrease extravasation rates for US-guided peripheral vascular access by providing guidance on catheter length selection.

DETAILED DESCRIPTION:
The purpose of this study is to compare catheter length and extravasation rates for US guided peripheral IV insertion in a subset of emergency department patients with difficult IV access. Physicians, Emergency RNs, and Emergency Technicians can be taught to use US guidance to start peripheral IV in the ED. The optimal length of catheter to use for this procedure is unknown. This study will provide data on the length of catheter required to minimize extravasation. There is no guideline on catheter length selection for US-guided peripheral vascular access. This study may decrease extravasation rates for US-guided peripheral vascular access by providing guidance on catheter length selection.

The study design is a randomized non-blinded clinical trial of extravasation rates of US guided peripheral vascular access related to intravenous catheter length and venous depth in the ED. Primary endpoint is duration of usable vascular access. Secondary endpoints are catheter length, venous depth, time of procedure, successful cannulation, reasons for failure, number of skin punctures, site of cannulation, sonographic technique, type of provider obtaining access and complications.

ELIGIBILITY:
Inclusion Criteria:

* two failed traditional IV attempts by a nurse
* need for IV access as determined by the treating physician
* age 18 and greater

Exclusion Criteria:

* less than age 18
* subjects needing a central venous catheter
* patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Extravasation rates | 48 hours
  compare catheter length and extravasation rates for US guided peripheral IV insertion in a subset of emergency department patients with difficult IV access

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sierzenski, MD, RDMS, Study Director — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States